CLINICAL TRIAL: NCT05492006
Title: Immune Response and Affective States of Elderly and 50+ Individuals After Intentional and Indirect Contact With Nature: a Randomized Controlled Clinical Trial
Brief Title: Immune Response and Affective States of Elderly and 50+ Individuals After Intentional and Indirect Contact With Nature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Paulo de Tarso Ricieri de Lima (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: e-Nature NK
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-03

CONDITIONS: Elderly
Keywords: health promotion; healthy aging; nature; immunological; older
MeSH Terms: interventions — Forest Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: intentional contact with nature (Active Comparator): Group A volunteers will take a light walk along the park with green space in a single 1-hour session with an emphasis on sense-directed appreciation guided by research team.
  Interventions: Behavioral: Intentional contact with nature
- Group B: indirect contact with nature (Active Comparator): The members of Group B will watch a video with the images of nature during 4 consecutive 15-minute sessions accompanied by the researcher, totaling 1 hour.
  Interventions: Behavioral: Indirect contact with nature

INTERVENTIONS:
Behavioral: Indirect contact with nature — The participants will watch a video with validated images of nature from e-Nature Positive Emotions Photography Database (e-NatPOEM). Four fifteen-minute sessions will be held on four consecutive days, totaling 1 hour.
  Other Names: e-NatPOEM
  Arms: Group B: indirect contact with nature
Behavioral: Intentional contact with nature — The participants will take a light walk in a park with green spaces guided by research team in a single 1-hour session, with an emphasis on sense-directed appreciation.
  Other Names: Forest Bathing
  Arms: Group A: intentional contact with nature

SUMMARY:
Randomized clinical trial on the influence of intentional and indirect contact with nature on the immune response and affective states in people aged 50 years or older.

DETAILED DESCRIPTION:
Interaction with nature creates a state of physical relaxation, helping the individual to manage stress and promote health. Along with the ability to reduce stress, nature has been shown to improve immune function in some specific environments. Science already proves that stress conditions affect the immune capacity, generating pathological immune responses and inflammatory responses inappropriate. Therefore, if contact with nature is capable of reducing stress, through this study can find manifestations of improvement of the functions immunological.

This clinical trial aims to analyze intentional (Forest Bathing) and indirect contact (e-NatPOEM) with nature. After informed consent form, participants will be randomized to the study arms. Will be evaluated cells and enzymes of the of the immune system and affective states immediately before the intervention, 30 minutes post intervention, and within 48 hours and four weeks after the intervention. The hypothesis of our study is that both nature-based interventions will stimulate the immune system and will improve affective states. However, intentional direct contact with nature will have superior results than indirect contact.

ELIGIBILITY:
Inclusion Criteria:

* individuals of both sexes
* capable of physical and mental to carry out the proposed activities
* capable of mental to fill in the questionnaires.

Exclusion Criteria:

* autoimmune diseases
* chronic or acute inflammatory diseases
* disease that affects the response of the immune system
* neuromuscular problems
* oncological diseases and neoplastic
* individuals being treated with immunosuppressive drugs or that affect the immune system
* individuals who are under the influence of alcohol or other substances that interfere with cognitive ability
* those who have had contact intentional relationship with nature in the 30-day period prior to participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Concentration of Cytokines in Soluble Immune Profile at 30 minutes post intervention, within 48 hours post intervention and within 4 weeks post intervention. | immediately pre intervention, 30 minutes post intervention, within 48 hours post intervention and within 4 weeks post intervention
  Quantify the change from baseline pre intervention in concentration of cytokines in plasma pg/ml (GM-CSF, IFNγ, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12 (p70), IL-3, IL-17A, IL-21, IL-23, ITAC, MIP-1α, MIP 1β, MIP -3 and TNF-α) in comparison the concentrations between the periods of 30 minutes post intervention, within 48 hours post intervention and within 4 weeks post intervention
Change from baseline percentage and absolute number levels of Cellular Immune Profile at 30 minutes post intervention, within 48 hours post intervention and within 4 weeks post intervention | immediately pre intervention, 30 minutes post intervention, within 48 hours post intervention and within 4 weeks post intervention.
  Quantify the changes from baseline pre intervention of frequencies in percentage of cells and absolute number in the blood of the subpopulation of lymphocytes and NK and their memory status within the period of 30 minutes post intervention, 48 hours and 4 weeks post intervention
Change from baseline percentage and absolute number levels of Cellular Immune Profile (others) at 30 minutes post intervention, within 48 hours and within 4 weeks post intervention | immediately pre intervention, 30 minutes post intervention, within 48 hours post intervention and within 4 weeks post intervention.
  To evaluate changes from baseline pre intervention of frequencies, percentage of cells positive for these biomarkers and intensity of expression in the pointed cells. Inhibiting, activating, effector and lytic molecules during the period of 30 minutes post intervention, within 48 hours and within 4 weeks post intervention.

SECONDARY OUTCOMES:
Change from baseline affective states at 30 minutes post intervention, within 48 hours post intervention and within 4 weeks post intervention. | immediately pre intervention, 30 minutes post intervention, within 48 hours post intervention and within 4 weeks post intervention.
  Will be applied the Profile of Mood States - POMS. It is one of the most used instruments in psychology to assess the states emotions and mood states, as well as the variation associated with them.
  Assesses six transient mood states: tension, depression, anger, vigor, fatigue and mental confusion. Each item can be rated on a Likert-type frequency scale of sensations, ranging from 0 (not at all) to 4 (extremely). Scores are not applicable to this scale.

CONTACTS AND LOCATIONS:
Overall Officials: Eliseth R Leão, PhD, Principal Investigator — Hospital Israelita Albert Einstein; Roberta M Savieto, MNP, Study Chair — Hospital Israelita Albert Einstein; Gabriela AG Gouveia, BPT, Study Chair — Beneficência Portuguesa de São Paulo
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dal Fabbro D, Catissi G, Borba G, Lima L, Hingst-Zaher E, Rosa J, Victor E, Bernardes L, Souza T, Leao E. e-Nature Positive Emotions Photography Database (e-NatPOEM): affectively rated nature images promoting positive emotions. Sci Rep. 2021 Jun 3;11(1):11696. doi: 10.1038/s41598-021-91013-9. PMID 34083616